CLINICAL TRIAL: NCT06272058
Title: Pharmacokinetics, Safety, and Tolerability of BI 685509 in Subjects With Severe Liver Impairment (Child-Pugh Classification C) as Compared to Healthy Subjects
Brief Title: A Study to Test How Avenciguat (BI 685509) is Taken up in the Body of People With and Without Liver Problems
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1366-0034
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Avenciguat (BI 685509) severe hepatic impairment (Child-Pugh C) (Experimental)
  Interventions: Drug: Avenciguat (BI 685509)
- Avenciguat (BI 685509) normal hepatic function (Experimental)
  Interventions: Drug: Avenciguat (BI 685509)

INTERVENTIONS:
Drug: Avenciguat (BI 685509) — Avenciguat (BI 685509)

SUMMARY:
This study is open to people with and without severe liver problems. People can join the study if they are 18 to 80 years of age and have a body mass index (BMI) between 18.5 and 42 kg/m2.

Avenciguat (BI 685509) is a medicine that is being developed to treat high blood pressure in the portal vein (main vessel going to the liver). The purpose of this study is to find out whether having liver problems influences how Avenciguat (BI 685509) is taken up in the body. All participants take Avenciguat (BI 685509) once as a tablet.

Participants are in the study for slightly longer than 1 month. Following the screening period of about 4 weeks, they stay at the study site for 4 nights. Afterwards, there are 2 visits to the study site. The site staff measures the amount of Avenciguat (BI 685509) in the blood. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 and ≤80 years at screening
* Body mass index (BMI) of 18.5 to 42 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Either male subject, or female subject who meet any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal), plus condom
  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
  * Sexually abstinent
  * A vasectomised sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant
  * Surgically sterilised (including hysterectomy)
  * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of Follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Applying only to participants with impaired hepatic function:

* Stable hepatic impairment (Child-Pugh score 10 - 15 point consistent with severe hepatic impairment) due to parenchymal liver disease, which is confirmed and documented by at least one of the following: medical history, physical examination, hepatic ultrasound, computed tomography (CT) scan, magnetic resonance imaging (MRI), and/or liver biopsy and defined as no clinically significant change in disease status within 4 weeks, as judged by the Investigator
* Absence of significant abnormalities, as based on a complete medical history including a full physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests at both screening and admission to trial site, with the exception of findings that in the opinion of the investigator are consistent with the participant's hepatic impairment.
* Medication and/or treatment regimens must have been stable (i.e., no dose adjustments) for at least 7 days or 5 half-lives whichever longer prior to the planned randomisation, and should be kept stable until study completion. Fluctuating treatment regimens may be considered for inclusion on a case-by-case basis if the underlying disease is under control in the opinion of the investigator and must be agreed to by both the investigator and the sponsor's medical monitor.

Applying only to healthy participants with normal hepatic function:

- Healthy subjects according to the assessment of the investigator (as based on a complete medical history including a physical examination, vital signs (BP, PR), 12- lead ECG, and clinical laboratory tests), and individually matched to participants with hepatic impairment according to sex, age and weight.

Exclusion Criteria:

* Any medical condition or finding in the medical examination that in the investigator's opinion assessed as clinically relevant, poses a safety risk for the subject or may interfere with the study objectives (except for conditions associated with hepatic impairment in subjects with compromised hepatic function)
* Repeated measurement of systolic blood pressure outside the range of 100 to 150 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 70 to 100 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any surgical or medical condition that may significantly interfere with the pharmacokinetics of the trial medication (eg, prior bariatric surgery, gastrectomy, ileal resection)
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin
* Intake of restricted concomitant therapy or any concomitant therapy considered likely (based on Investigator judgement) to interfere with the safe conduct or may influence the primary and/or secondary endpoints of the trial within 30 days or 5 half-lives whichever longer prior to planned administration of the trial medication.
* Ongoing chronic alcohol or drug use, that in the investigator's opinion, makes the patient an unreliable trial participant or unlikely to complete the trial.

Further exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-05-03 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 6 days
Maximum measured concentration of the analyte in plasma (Cmax) | up to 6 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 6 days
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to 6 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com